CLINICAL TRIAL: NCT04948749
Title: Drug Eluting Stenting and Aggressive Medical Treatment for Preventing Recurrent Stroke in Intracranial Atherosclerotic Disease Trial: a Prospective, Randomized, Open-labelled, Blinded End-point Trial (DREAM-PRIDE)
Brief Title: Drug Eluting Stenting and Aggressive Medical Treatment for Preventing Recurrent Stroke in Intracranial Atherosclerotic Disease Trial
Acronym: DREAM-PRIDE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HX-A-018(2021)
Record Dates: First submitted 2021-06-16; First posted 2021-07-02 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: ICAD - Intracranial Atherosclerotic Disease; ICAS - Intracranial Atherosclerosis; Drug-eluting Stent; Stroke; Drug Eluting Stents (DES); Medical Treatment
Keywords: Stroke; Drug-eluting stent; Medical treatment; ICAD-Intracranial Atherosclerotic Disease; ICAS-Intracranial Atherosclerosis; Drug Eluting Stents (DES)
MeSH Terms: conditions — Intracranial Arteriosclerosis; Stroke | interventions — Risk Factors

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Drug-eluting stent implantation with aggressive medical treatment group (Experimental): DES implantation (The Maurora ® Sirolimus Eluting Stent System) combined with aggressive medical treatment (aspirin 100 mg per day for the entire follow-up, clopidogrel 75 mg per day, or ticagrelor 90 mg twice per day for 6 months); management of risk factors (hypertension, diabetes, lipoprotein metabolism disorder, smoking and exercise)
  Interventions: Device: Drug Eluting Stent implantation; Drug: Aggressive medical treatment; Behavioral: Risk factor management
- Standard medical treatment group (Active Comparator): Standard medical treatment (aspirin 100 mg per day for the entire follow-up, clopidogrel 75 mg per day, or ticagrelor 90 mg twice per day for 3 months after enrolment), management of risk factors (hypertension, diabetes, lipoprotein metabolism disorder, smoking and exercise)
  Interventions: Behavioral: Risk factor management; Drug: Standard medical treatment

INTERVENTIONS:
Device: Drug Eluting Stent implantation — The Maurora ® Sirolimus Eluting Stent System for intracranial PTA treatment comprises of a balloon expandable sirolimus eluting stent and a delivery catheter that features a rapid exchange catheter design with a semi-compliant balloon located at its distal end.
  Other Names: Maurora ® Sirolimus Eluting Stent implantation
  Arms: Drug-eluting stent implantation with aggressive medical treatment group
Drug: Aggressive medical treatment — Aggressive medical treatment consists of dual antiplatelet treatment (aspirin 100 mg per day for the entire follow-up, clopidogrel 75 per day mg, or ticagrelor 90 mg twice per day for 6 months after enrollment).
  Other Names: Dual antiplatelet therapy for 6 months
  Arms: Drug-eluting stent implantation with aggressive medical treatment group
Behavioral: Risk factor management — Management of risk factors (hypertension, diabetes, lipoprotein metabolism disorder, smoking and exercise)
  Other Names: Risk factor and life style management
Drug: Standard medical treatment — Standard medical treatment consists of dual antiplatelet treatment (aspirin 100 mg per day for the entire follow-up, clopidogrel 75 per day mg, or ticagrelor 90 mg twice per day for 3 months after enrollment).
  Other Names: Dual antiplatelet therapy for 3 months
  Arms: Standard medical treatment group

SUMMARY:
The aim of DREAM-PRIDE is to evaluate whether implantation of drug-eluting stent (DES) combined with aggressive medical treatment is more efficacious in prevention of 1-year stroke recurrence than standard medical treatment alone for symptomatic intracranial atherosclerotic disease.

DETAILED DESCRIPTION:
This trial is a prospective, multi-center, 1:1 randomized using drug-eluting (Sirolimus) stent combined with aggressive medical treatment versus standard medical treatment to treat symptomatic intracranial atherosclerotic disease. Primary efficacy endpoints (any of the following): 1) any stroke or death within 30 days after enrollment, 2) any stroke or death within 30 days after a revascularization procedure of the qualifying lesion during follow-up, 3) ischemic stroke in the territory of the qualifying artery beyond 30 days to 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 85 years
2. Patients with ischemic stroke within 30 days of enrolment attributed to 70% to 99% stenosis of a major intracranial artery (internal carotid artery [C4-C7], middle cerebral artery [M1], vertebral artery [V4], or basilar artery) on CTA (According to WASID method)
3. The diameter of the target vessel between 2.0mm - 4.5mm
4. The stenosis lesion length ≤ 14 mm
5. Baseline modified Rankin Scale (mRS) score ≤ 3
6. Patient understands the purpose and requirements of the study, and has provided informed consent

Exclusion Criteria:

1. Ischemic stroke occurred within 7 days before enrolment
2. Tandem extracranial or intracranial stenosis (70%-99%) or occlusion that is proximal or distal to the target intracranial lesion (NOTE: an exception is allowed if stenosis or occlusion involves a single vertebral artery proximal to a symptomatic basilar artery stenosis and the contralateral vertebral artery is supplying the basilar artery)
3. Bilateral intracranial vertebral artery stenosis of 70%-99% and uncertainty about which artery is symptomatic (NOTE: an exception is that if bilateral vertebral arteries with 70%-99% stenosis but unequal in size, the dominant side is considered as symptomatic)
4. Unilateral vertebral artery stenosis of 70%-99% with normal contralateral vertebral artery
5. Stroke caused by perforating artery occlusion
6. CT angiographic evidence of severe calcification at target lesion
7. Any history of brain parenchymal or subarachnoid, subdural or extradural haemorrhage in the past 6 weeks
8. Intracranial artery stenosis caused by non-atherosclerotic lesions, including: arterial dissection, Moyamoya disease, vasculitis disease, herpes zoster, varicella-zoster or other viral vascular diseases, neurosyphilis, any other intracranial infections, any intracranial stenosis related to cerebrospinal fluid cells, radiation-induced vascular disease, fibromuscular dysplasia, sickle cell disease, neurofibromatosis, central nervous system benign vascular disease, postpartum vascular disease, suspected vasospasm, suspicious embolism recanalization, etc
9. History of stenting of an intracranial artery
10. Presence of any unequivocal cardiac source of embolism
11. Combined with intracranial tumor, aneurysm or intracranial arteriovenous malformation
12. Cannot tolerate dual antiplatelet therapy
13. Contraindications to heparin, rapamycin, contrast and local or general anesthesia
14. Hemoglobin<100g/L, platelet count <100×109/L
15. Severe hepatic and renal dysfunction
16. INR>1.5 or there are uncorrectable factors leading to bleeding
17. Major surgery within the past 30 days or planned within 90 days
18. Renal artery, iliac artery, and coronary artery requiring simultaneous intervention
19. Life expectancy <1 year
20. Pregnant or lactating women
21. Cannot complete the follow-up due to cognitive, emotional or mental illness
22. Other situations that are not suitable for enrolment according to the judgement of the investigator
23. Enrolment in another study that would conflict with the current study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 792 (Estimated)
Dates: Start 2021-07-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Any stroke or death within 30 days of enrollment or any revascularization procedure OR an ischemic stroke in the territory of the symptomatic intracranial artery between 31 day to 1 year. | 12 months after enrollment
  Primary endpoints are composite event of (1) any stroke or death within 30 days after enrollment, (2) any stroke or death within 30 days after revascularization procedure of the qualifying lesion during follow-up, and (3) ischemic stroke in the territory of the qualifying artery from 31 days to 1 year. Ischemic stroke is defined as a new focal neurological deficit of sudden onset, that is associated with infarction lesion on CT or MRI. Ischemic strokes are classified as in or out of the territory of the symptomatic intracranial artery. Symptomatic brain hemorrhage is defined as parenchymal, subarachnoid, or intraventricular hemorrhage detected by CT or MRI that is associated with new neurological signs or symptoms (headache, change in level of consciousness, focal neurological symptoms) lasting ≥ 24 hours or a seizure.
Severe or moderate bleeding (GUSTO score) | 12 months after enrollment
  Bleeding events were defined according to the Global Use of Strategies to Open Occluded Coronary Arteries (GUSTO) classification for severe or life-threatening, moderate, or mild bleeding:
  Severe or life-threatening- Either intracranial hemorrhage or bleeding that causes hemodynamic compromise and requires intervention
  Moderate- Bleeding that requires blood transfusion but does not result in hemodynamic compromise
  Mild- Bleeding that does not meet criteria for either severe/life-threatening or moderate bleeding

SECONDARY OUTCOMES:
Residual stenosis after the procedure in DES group | At the end of the procedure
  Degree of residual stenosis was measured and calculated according to the methods of the Warfarin-Aspirin Symptomatic Intracranial Disease (WASID) trial.
In-stent restenosis (ISR) rate in DES group within 12 months | 12 months after enrollment
  The ISR is defined as >50% stenosis within or immediately adjacent (within 5 mm) of the implanted stent and >20% absolute luminal loss.
Disabling stroke within 1 year | 12 months after enrollment
  defined as modified Rankin Scale > 3 at 1 year visit
Any stroke, death or myocardial infarction within 1 year | 12 months after enrollment
  Any stroke included ischemic stroke and symptomatic brain hemorrhage. Symptomatic brain hemorrhage refers to parenchymal, subarachnoid, or intraventricular hemorrhage that was associated with a seizure or with symptoms or signs lasting 24 hours or longer.
Major non-stroke hemorrhage within 1 year | 12 months after enrollment
  A major non-stroke-related hemorrhage was defined as any subdural or epidural hemorrhage or a systemic hemorrhage requiring hospitalization, blood transfusion, or surgery.
Modified Rankin Scale score at 1 year | 12 months after enrollment
  The range of modified Rankin Scale was from 0 to 6. 0-No symptoms;1-No significant disability;2-Slight disability;3-Moderate disability;4-Moderately severe disability;5-Severe disability;6 -Dead.A higher score indicates worse a outcome.
Death within 1 year | 12 months after enrollment
  Death within 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yongjun Wang, MD, Principal Investigator — Beijing Tiantan Hospital; Zhongrong Miao, MD, Principal Investigator — Beijing Tiantan Hospital
Locations (18):
- China (18):
  - Beijing Tiantan Hospital, Beijing, Beijing Municipality
  - Beijing Daxing District People's Hospital, Beijing, Beijing Municipality
  - Hejian People's Hospital, Cangzhou, Hebei
  - North China University of Science and Technology Affiliated Hospital, Tangshan, Hebei
  - Xingtai City Third Hospital, Xingtai, Hebei
  - General Hospital of The Yangtze River Shipping, Wuhan, Hubei
  - Baotou Central Hospital, Baotou, Inner Mongolia
  - Inner Mongolia Autonomous Region People's Hospital, Hohhot, Inner Mongolia
  - Tongliao City Hospital, Tongliao, Inner Mongolia
  - Wuhai People's Hospital, Wuhai, Inner Mongolia
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - The Second Norman Bethune Hospital of JilinUniversity,, Changchun, Jilin
  - General Hospital of Benxi Iron and Steel Co, Benxi, Liaoning
  - Shanxi Cardiovascular Hospital, Taiyuan, Shanxi
  - Shanxi Provincial People's Hospital, Taiyuan, Shanxi
  - The First Affiliated Hospital of College of Medicine, Hangzhou, Zhejiang
  - Lishui People's Hospital, Lishui, Zhejiang
  - Beilun People's Hospital of Ningbo City, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhou M, Wang H, Zeng X, Yin P, Zhu J, Chen W, Li X, Wang L, Wang L, Liu Y, Liu J, Zhang M, Qi J, Yu S, Afshin A, Gakidou E, Glenn S, Krish VS, Miller-Petrie MK, Mountjoy-Venning WC, Mullany EC, Redford SB, Liu H, Naghavi M, Hay SI, Wang L, Murray CJL, Liang X. Mortality, morbidity, and risk factors in China and its provinces, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2019 Sep 28;394(10204):1145-1158. doi: 10.1016/S0140-6736(19)30427-1. Epub 2019 Jun 24. PMID 31248666
- [Background] GBD 2016 Stroke Collaborators. Global, regional, and national burden of stroke, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet Neurol. 2019 May;18(5):439-458. doi: 10.1016/S1474-4422(19)30034-1. Epub 2019 Mar 11. PMID 30871944
- [Background] Chimowitz MI, Lynn MJ, Howlett-Smith H, Stern BJ, Hertzberg VS, Frankel MR, Levine SR, Chaturvedi S, Kasner SE, Benesch CG, Sila CA, Jovin TG, Romano JG; Warfarin-Aspirin Symptomatic Intracranial Disease Trial Investigators. Comparison of warfarin and aspirin for symptomatic intracranial arterial stenosis. N Engl J Med. 2005 Mar 31;352(13):1305-16. doi: 10.1056/NEJMoa043033. PMID 15800226
- [Background] Chimowitz MI, Lynn MJ, Derdeyn CP, Turan TN, Fiorella D, Lane BF, Janis LS, Lutsep HL, Barnwell SL, Waters MF, Hoh BL, Hourihane JM, Levy EI, Alexandrov AV, Harrigan MR, Chiu D, Klucznik RP, Clark JM, McDougall CG, Johnson MD, Pride GL Jr, Torbey MT, Zaidat OO, Rumboldt Z, Cloft HJ; SAMMPRIS Trial Investigators. Stenting versus aggressive medical therapy for intracranial arterial stenosis. N Engl J Med. 2011 Sep 15;365(11):993-1003. doi: 10.1056/NEJMoa1105335. Epub 2011 Sep 7. PMID 21899409
- [Background] Shin YS, Kim BM, Suh SH, Jeon P, Kim DJ, Kim DI, Kim BS, Kim KH, Heo JH, Nam HS, Kim YD. Wingspan stenting for intracranial atherosclerotic stenosis: clinical outcomes and risk factors for in-stent restenosis. Neurosurgery. 2013 Apr;72(4):596-604; discussion 604. doi: 10.1227/NEU.0b013e3182846e09. PMID 23277374
- [Background] Jin M, Fu X, Wei Y, Du B, Xu XT, Jiang WJ. Higher risk of recurrent ischemic events in patients with intracranial in-stent restenosis. Stroke. 2013 Nov;44(11):2990-4. doi: 10.1161/STROKEAHA.113.001824. Epub 2013 Aug 20. PMID 23963335
- [Background] Lu WD, Huang CW, Li YH, Chen JY. Multiple Mechanisms in 1 In-Stent Restenosis Assessed by Optical Coherence Tomography. JACC Cardiovasc Interv. 2017 Nov 27;10(22):2340-2341. doi: 10.1016/j.jcin.2017.07.017. Epub 2017 Nov 1. No abstract available. PMID 29102578